CLINICAL TRIAL: NCT04017117
Title: Comparative Study Between Custom-made Polyether Ether Ketone and Titanium Mesh for Augmentation of Atrophic Posterior Mandible. Randomized Clinical Trial
Brief Title: Augmentation of Atrophic Mandibule Using Poly Ether Ether Ketone Mesh
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adham Zakaria, Master Degree Candidate., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-06-19
Record Dates: First submitted 2019-06-25; First posted 2019-07-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Mandible Small
MeSH Terms: conditions — Micrognathism

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial. A trial will be carried out in hospital of Oral and Maxillofacial surgery department,Faculty of Oral and Dental Medicine Cairo University Equal randomization parallel group study positive controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom Made Poly Ether Ether Ketone Mesh (Experimental): Applying Poly Ether Ether Ketone mesh with mix of autogenous bone graft and bone substitute in posterior atrophic mandible for augmentation
  Interventions: Procedure: under local anasthesia,Ridge Augmention of posterior atrophic mandible by using mix of autogenous bone graft and bone substitutes is used under PEEK mesh
- Conventional Titanium mesh (Active Comparator): Applying Titanium mesh with mix of autogenous bone graft and bone substitute in posterior atrophic mandible for augmentation
  Interventions: Procedure: under local anasthesia,Ridge Augmention of posterior atrophic mandible by using mix of autogenous bone graft and bone substitutes is used under PEEK mesh

INTERVENTIONS:
Procedure: under local anasthesia,Ridge Augmention of posterior atrophic mandible by using mix of autogenous bone graft and bone substitutes is used under PEEK mesh — comparing between PEEK mesh and Titanium mesh for augmentation of posterior atrophic mandible using mix of autogenous bone graft and bone substitute.

SUMMARY:
Comparative study between custom-made polyether ether ketone and titanium mesh for augmentation of atrophic posterior mandible.

DETAILED DESCRIPTION:
Designing and manufacturing

1. The CBCT images of the patient will be used to build a digital model using a 3D planning software (Mimics innovation suite). Based on this model, a machine will be used to mill a pressed and pre-sintered body of PEEK to the desired macroscopic shape.

2. The size of the machined sheet is enlarged in order to compensate for the sintering shrinkage performed at 1450 C.

3. After manufacturing, the sheet will be cleaned in an ultrasonic bath of 70% alcohol for 15 min, followed by a brief heating to 1200 C.

4. It will be again cleaned in an ultrasonic bath for 3x15 min using 90% alcohol.

5. Thereafter the sheet was placed in an autoclave and sterilized using a standard program.

6. The sheets will have a thickness of approximately 0.5 - 0.7 mm. b. Surgery

1. The intraoral area is initially cleaned with chlorhexidine 1 mg/ml.
2. Local anesthesia is administered.
3. Horizontal crestal incisions are made lingual of the mid-crest within the keratinized tissue. Vertical releasing incisions are placed on the buccal aspect of the surgical site in the usual manner to provide adequate access and to allow for eventual coronal repositioning.
4. Then, a full-thickness mucoperiosteal flap is reflected to completely expose the atrophic ridge.
5. The cortex of the mandibular crest is generously perforated to produce bleeding in multiple sites. The pilot holes for the fixation screws were also prepared at this time.
6. The barrier is inserted over the mandible and compressed into place, the fixation screws are inserted and no adaptation will be needed as the barrier is custom-made for the edentulous ridge.
7. The ceramic sheets is cleaned with 3% hydrogen peroxide prior to soft tissue closure.
8. After fixation of the sheets, the buccal flaps should be coronally repositioned.
9. Split-thickness periosteal releasing incisions are completed to aid in primary tension-free closure. The flap margins are then advanced over the barrier and approximated to evaluate for tension-free closure.
10. After a mean of 6 months of uneventful healing, the augmented sites are reopened. The ceramic barrier and fixation screws are identified and removed, followed by Dental implant.

Post-operative care:

Avoid traumatization of the surgical site. Patients must abstain from brushing at the surgical area. Instead, a disinfecting mouth rinse should be used (e.g. chlorhexidine 0.2%).

Instruct the patient not to touch or manipulate the surgical area. Ice packs for 10 minutes every 30 minutes for 24 hours. Do not use removable dentures during the expansion phase. Temporary fixed partial dentures must be adjusted to the expected tissue gain.

No consume of tobacco

Post-operative medications will be prescribed as follows:

Amoxicillin/clavulanic acid tablets 10mg/kg every 12 hours for 7 days, diclofenac potassium 50mg every 8 hours for 4 days and then as needed, metronidazole 5 mg/kg every 8 hours for 7 days and chlorhexidine gluconate 0.1% mouthwash 3 times daily for 14 days.

11b. Criteria for discontinuing or modifying intervention: No protocol for discontinuation of the procedure. 11c. Strategies to improve adherence to intervention: Face to face adherence reminder session will take place to stress on the post-operative instructions at the following time intervals.

Patients were recalled every other day to monitor soft tissue healing for the first week, one visit weekly for the first month then monthly for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with atrophic posterior mandible
2. Both sexes
3. No intraoral soft and hard tissue pathology
4. No systemic condition that contraindicate implant placement

Exclusion Criteria:

1. Untreated gingivitis, periodontitis
2. Insufficient oral hygiene
3. Previous radiation therapy the head and neck neoplasia, or bone augmentation to implant site.
4. Systemic disorders
5. Heavy smoking more than 20 cigarettes per day
6. Bone pathology
7. Psychiatric problems
8. Emotional instability
9. Unrealistic aesthetic demands

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-11-25 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Vertical amount of bone increased (length in millimeters). horizontal amount f bone increased after augmentation (width in millimeters). | 6 months
  Length (Vertical Augmentation) Width (horizontal augmentation) gained after augmentation of atrophic mandible in millimeters using cone beam computed tomography (measuring tool) measurment tools : with the aid of cone beam computed tomography

SECONDARY OUTCOMES:
Rate of Soft Tissue Dehiscence | 6 months
  which mesh will cause soft tissue dehiscence more.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Shehab, PHD, Study Director — Professor of Oral and Maxillofacial Surgery - Cairo University.; Khaled A Salaheddin, PHD, Study Director — Lecturer of Oral and Maxillofacial Surgery - Cairo University.
Locations (1):
- Faculty Of Dental and Oral Medicine-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misch CM. Bone augmentation of the atrophic posterior mandible for dental implants using rhBMP-2 and titanium mesh: clinical technique and early results. Int J Periodontics Restorative Dent. 2011 Nov-Dec;31(6):581-9. PMID 22140660
- [Background] Her S, Kang T, Fien MJ. Titanium mesh as an alternative to a membrane for ridge augmentation. J Oral Maxillofac Surg. 2012 Apr;70(4):803-10. doi: 10.1016/j.joms.2011.11.017. Epub 2012 Jan 28. PMID 22285340
- [Result] Pieri F, Corinaldesi G, Fini M, Aldini NN, Giardino R, Marchetti C. Alveolar ridge augmentation with titanium mesh and a combination of autogenous bone and anorganic bovine bone: a 2-year prospective study. J Periodontol. 2008 Nov;79(11):2093-103. doi: 10.1902/jop.2008.080061. PMID 18980518
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18980518
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22140660
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/22285340